CLINICAL TRIAL: NCT02715128
Title: Disorder-tailored Transcranial Direct Current Stimulation (tDCS) of the Prefrontal Cortex: fMRI Study in Major Depression and Schizophrenia
Brief Title: Disorder-tailored Transcranial Direct Current Stimulation (tDCS) of the Prefrontal Cortex
Acronym: MRSDC1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Daniel Keeser, Dr. rer. biol. hum., Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 493-14
Record Dates: First submitted 2016-03-16; First posted 2016-03-22 (Estimated); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Major Depressive Disorder; Schizophrenia
MeSH Terms: conditions — Depressive Disorder, Major; Schizophrenia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- real tDCS (Active Comparator): anode over electrode position F3, cathode over F4, 20 min, 2mA intensity
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- sham tDCS (Sham Comparator): frequency and duration correspondent active tDCS, ramp in and ramp out periods only without intermittent stimulation
  Interventions: Device: Transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — non-invasive electric brain stimulation method

SUMMARY:
Major depressive disorder (MDD) is a common, recurrent, and frequent chronic disorder. Among others, deficient cognitive control over emotional distraction is a central characteristic of MDD (Ochsner & Gross 2005; Disner et al. 2011; Beck 2008). Hypoactivation of the dorsolateral prefrontal cortex (DLPFC) has been linked with this deficit (Dolcos & McCarthy 2006). Moreover, aberrant functional connectivity patterns have been found in MDD patients (Kaiser et al. 2015). Transcranial direct current stimulation (tDCS) is a non-invasive brain stimulation method that has been largely investigated in experimental neurosciences and tDCS of the prefrontal cortex (PFC) has been proposed as novel treatment in MDD. In addition, it is increasingly investigated as treatment for negative symptoms in schizophrenia (SCZ) (Brunelin et al. 2012). So far, prefrontal tDCS has been shown to enhance cognitive control over emotional distraction in MDD patients (Wokenstein & Plewnia 2013). Also, tDCS-induced connectivity changes found in fMRI studies comparing resting-state networks configurations before and after prefrontal tDCS may reflect a state of enhanced alertness (Keeser, Meindl, et al., 2011; Park et al., 2013).

The aim of this study is to investigate the neurophysiological correlates of tDCS effects in patients with different psychiatric disorders for which tDCS is a possible intervention, in particular MDD and SCZ, as compared to healthy individuals. For this purpose, we determine the most promising protocol in from investigations in healthy volunteers and apply this protocol in the patient sample including age- and gender-matched controls. First, functional magnetic resonance imaging (fMRI) data is collected during the execution of a cognitive control task as well as during a resting-state condition together with application of real or sham tDCS inside the scanner. It is hypothesized that prefrontal tDCS as compared to sham a) reduces distractibility by compensating for deficient DLPFC activity and b) enhances functional connectivity in networks associated with externally directed attention or cognitive engagement. Second, magnetic resonance spectroscopy (MRS) is performed to measure concentrations of GABA and glutamate in target regions of tDCS. It is hypothesized that tDCS effects are mediated via modulation of the inhibitory/excitatory systems and GABA and glutamate are used as markers of these systems.

In this placebo-controlled study healthy volunteers and patients with a diagnosis of MDD or SCZ receive a single treatment with prefrontal tDCS (anode over electrode position F3, cathode over F4, 20 min, 2mA intensity) or sham tDCS (frequency and duration correspondent active tDCS, ramp in and ramp out periods only without intermittent stimulation). We conduct resting-state and MRS measurements combined with application of tDCS in the fMRI scanner. Subsequently, participants perform the cognitive control task (in dependence of Plewnia, C., Schroeder, P. A., & Wolkenstein, L. (2015)) in the scanner. The participants are assigned to either the real or sham tDCS condition according to a randomised, double-blind parallel design.

ELIGIBILITY:
Inclusion Criteria:

* Men and women 18-60 years of age.
* Capable and willing to provide informed consent.
* MDD: Primary ICD-10 diagnosis of Major Depression and a total HDRS-21 ≥15 and/or BDI ≥15 at the screening visit; no antidepressant medication and stable medication ≥4 days before study onset and during study period.
* SCZ: Primary ICD10 diagnosis of Schizophrenia and a stable antipsychotic medication ≥1 weeks before study onset and during study period.

Exclusion Criteria:

* Contraindications for brain stimulation, such as history of brain surgery or severe brain injury, as well as contraindications for MRI, such as metallic implants, any other non-MR safe implants, or claustrophobia.
* Investigators, site personnel directly affiliated with this study, and their immediate families (immediate family is defined as a spouse, parent, child or sibling, whether by birth or legal adoption).
* Acute risk for suicide (MADRS, item 10 score of >4 or as assessed by the C-SSRS, agree to item 4 and/or agree to item 5).
* Treatment with electroconvulsive therapy in the present episode.
* Treatment with deep brain stimulation or vagus nerve stimulation and/or any other intracranial implants (clips, cochlear implants).
* Any other relevant psychiatric axis-I- and/or axis-II-disorder.
* Any relevant instable medical condition.
* Pregnancy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-03 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
FMRI modulations | 2 hours
  differences in the cognitive control task (performance and activations) between the sham and real group as well as changes in resting-state connectivity between and within (following stimulation compared to baseline) groups
GABA and Glutamate modulations | 2 hours
  differences in excitatory and inhibitory system modulation visualised via GABA and Glutamate concentrations determined by H1-MRS measurements

SECONDARY OUTCOMES:
Clinical trajectories | 8 weeks
  Influence of observed online modulatory effects on clinical trajectories in patients

CONTACTS AND LOCATIONS:
Overall Officials: Frank Padberg, Prof. Dr., Principal Investigator — Ludwig-Maximilians-Universität München
Locations (1):
- Department of Psychiatry and Psychotherapy, Ludwig-Maximilian University Munich, Munich, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Keeser D, Meindl T, Bor J, Palm U, Pogarell O, Mulert C, Brunelin J, Moller HJ, Reiser M, Padberg F. Prefrontal transcranial direct current stimulation changes connectivity of resting-state networks during fMRI. J Neurosci. 2011 Oct 26;31(43):15284-93. doi: 10.1523/JNEUROSCI.0542-11.2011. PMID 22031874
- [Background] Park CH, Chang WH, Park JY, Shin YI, Kim ST, Kim YH. Transcranial direct current stimulation increases resting state interhemispheric connectivity. Neurosci Lett. 2013 Feb 28;539:7-10. doi: 10.1016/j.neulet.2013.01.047. Epub 2013 Feb 13. PMID 23416318
- [Background] Kaiser RH, Andrews-Hanna JR, Wager TD, Pizzagalli DA. Large-Scale Network Dysfunction in Major Depressive Disorder: A Meta-analysis of Resting-State Functional Connectivity. JAMA Psychiatry. 2015 Jun;72(6):603-11. doi: 10.1001/jamapsychiatry.2015.0071. PMID 25785575
- [Background] Ochsner KN, Gross JJ. The cognitive control of emotion. Trends Cogn Sci. 2005 May;9(5):242-9. doi: 10.1016/j.tics.2005.03.010. PMID 15866151
- [Background] Disner SG, Beevers CG, Haigh EA, Beck AT. Neural mechanisms of the cognitive model of depression. Nat Rev Neurosci. 2011 Jul 6;12(8):467-77. doi: 10.1038/nrn3027. PMID 21731066
- [Background] Beck AT. The evolution of the cognitive model of depression and its neurobiological correlates. Am J Psychiatry. 2008 Aug;165(8):969-77. doi: 10.1176/appi.ajp.2008.08050721. Epub 2008 Jul 15. PMID 18628348
- [Background] Dolcos F, McCarthy G. Brain systems mediating cognitive interference by emotional distraction. J Neurosci. 2006 Feb 15;26(7):2072-9. doi: 10.1523/JNEUROSCI.5042-05.2006. PMID 16481440
- [Background] Wolkenstein L, Plewnia C. Amelioration of cognitive control in depression by transcranial direct current stimulation. Biol Psychiatry. 2013 Apr 1;73(7):646-51. doi: 10.1016/j.biopsych.2012.10.010. Epub 2012 Dec 6. PMID 23219367
- [Background] Plewnia C, Schroeder PA, Wolkenstein L. Targeting the biased brain: non-invasive brain stimulation to ameliorate cognitive control. Lancet Psychiatry. 2015 Apr;2(4):351-6. doi: 10.1016/S2215-0366(15)00056-5. Epub 2015 Mar 31. PMID 26360088
- [Background] Brunelin J, Mondino M, Gassab L, Haesebaert F, Gaha L, Suaud-Chagny MF, Saoud M, Mechri A, Poulet E. Examining transcranial direct-current stimulation (tDCS) as a treatment for hallucinations in schizophrenia. Am J Psychiatry. 2012 Jul;169(7):719-24. doi: 10.1176/appi.ajp.2012.11071091. PMID 22581236
- See also: Related Info — http://gcbs.network/gcbs/projects/human-models/Work-Package-5.html